CLINICAL TRIAL: NCT02800850
Title: Bright Light Therapy for Individuals With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radford University (Other)
Collaborators: Commonwealth Care of Roanoke, Inc. (Unknown); Virginia Center on Aging (ARDRAF) (Unknown)
Responsible Party: Principal Investigator, Lisa L. Onega, Professor of Nursing, Radford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RadfordU
Record Dates: First submitted 2016-05-31; First posted 2016-06-15 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Dementia
Keywords: Dementia; Depression; Agitation; Bright Light
MeSH Terms: conditions — Dementia; Depression; Psychomotor Agitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bright Light Group (Experimental): Bright Light Exposure
  Interventions: Behavioral: Bright Light
- Control Group (Placebo Comparator): Placebo Light Exposure
  Interventions: Behavioral: Placebo Light

INTERVENTIONS:
Behavioral: Bright Light
  Arms: Bright Light Group
Behavioral: Placebo Light
  Arms: Control Group

SUMMARY:
Many older adults with dementia living in long-term care facilities experience depression and agitation, which cause angst and personal suffering. Prior to this research, evidence was inconclusive but indicated that bright light exposure may reduce depression and agitation in long-term care residents with dementia. The purpose of this study was to determine if the degree of improvement in depression and agitation scores over the course of eight weeks was significantly greater in persons with dementia receiving bright light exposure than in persons with dementia receiving placebo light exposure. Sixty individuals participated in the study, with 30 in the bright light group and 30 in the low level light group.

ELIGIBILITY:
Inclusion criteria were age 60 or older; diagnosis of dementia; ophthalmology screening indicating that the individual was able to perceive light and did not have cataracts, glaucoma, macular degeneration, or retinal problems; able to sit up and keep eyes open; and not too restless to sit for 30 minutes.

Exclusion criteria were age 59 or younger; no diagnosis of dementia; presence of cataracts, glaucoma, macular degeneration, or retinal problems; unable to sit up and keep eyes open; and too restless to sit for 30 minutes.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Depressive Symptom Assessment for Older Adults | After the eight-week experiment
Cohen-Mansfield Agitation Inventory (Frequency) | After the eight-week experiment

CONTACTS AND LOCATIONS:
Overall Officials: Lisa L Onega, PhD, RN, MBA, Principal Investigator — Radford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Onega LL, Pierce TW, Epperly L. Effect of Bright Light Exposure on Depression and Agitation in Older Adults with Dementia. Issues Ment Health Nurs. 2016 Sep;37(9):660-667. doi: 10.1080/01612840.2016.1183736. Epub 2016 Jun 2. PMID 27254531